CLINICAL TRIAL: NCT05523115
Title: An Exploratory Investigation of a Supplement to Promote Cognitive Health Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heights (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20250
Record Dates: First submitted 2022-08-26; First posted 2022-08-31 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Anxiety; Stress; Memory Deficits; Cortisol Overproduction
Keywords: memory; stress; anxiety; mood; focus
MeSH Terms: conditions — Anxiety Disorders; Memory Disorders; ACTH Syndrome, Ectopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heights Smart Supplement (Experimental): Participants will take the supplement over a 12 week period. There will be both biomarker outcomes and subjective outcomes reported by the participants via questionnaires.
  Interventions: Dietary Supplement: Heights Smart Supplement

INTERVENTIONS:
Dietary Supplement: Heights Smart Supplement — The ingredient list of the product includes the following:
  Algae oil Blueberry Extract Methylcobalamin (Vitamin B12) Cholecalciferol (Vitamin D3) Ascorbic acid (Vitamin C) Retinol acetate (Vitamin A) Calcium L-methylfolate (Folic Acid) D-biotin Pyridoxine hydrochloride (Vitamin B6) Calcium pantothenate (Vitamin B5) Nicotinamide (Vitamin B3) Riboflavin (Vitamin B2) Thiamine hydrochloride (Vitamin B1) D-Alpha tocopheryl acetate (Vitamin E) Chromium picolinate Potassium iodide Iron Citrate Sodium selenite Zinc citrate

SUMMARY:
The Smart Supplement has 20 vitamins and minerals that have strong track records of demonstrating positive health effects, both physiologically and cognitively. This twelve-week trial will examine the effectiveness and efficacy of Heights Smart Supplement on both biomarkers and subjective experiences from participants.

ELIGIBILITY:
Inclusion Criteria:

* In good general health with no major chronic conditions
* Must experience one of the following issues: brain fog
* OR issues with fatigue,
* OR sleep issues,
* OR trouble with focus and concentration,
* OR lead a busy, stressful life.
* Must have a fitness tracker that they use to track sleep behaviors.
* May be on a vegan/vegetarian diet

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Anyone currently taking other supplements focused on brain health, or multi vitamins, including additional iron supplements
* Anyone taking Thyroxine and Levothyroxine
* Anyone taking antidepressants (such as Sertraline or SSRIs like fluoxetine)
* Anyone on hormone replacement therapy
* Anyone taking blood pressure medication (such as linosipril)
* Anyone with a known allergic reaction
* Any chronic conditions, including oncological and psychiatric disorders

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in Measures of C-reactive protein | 12 weeks
  Biomarkers measured by a third party lab through blood samples submitted by participants.
Changes in Measures of cortisol | 12 weeks
  Biomarkers measured by a third party lab through blood samples submitted by participants.
Changes in Sleep Quality as measured via Fitness trackers and Questionnaires | 12 weeks
  Measurements taken via existing smart watches and report that data on the questionnaires.

SECONDARY OUTCOMES:
examine the subjective experiences of participants taking the Heights Smart Supplement. | 12 weeks
  The questionnaires for this study are specifically designed to understand changes in focus, anxiety embedded in mood & stress, memory, and overall well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hill, PhD, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided